CLINICAL TRIAL: NCT03101111
Title: Phase 2 Study of a Live Attenuated Measles Virus-Vectored Chikungunya Vaccine in a Previously Epidemic Area
Brief Title: Study of a Live Attenuated Chikungunya Vaccine in a Previously Epidemic Area
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Themis Bioscience GmbH (Industry)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MV-CHIK-204
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Results first posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2018-09

CONDITIONS: Chikungunya
MeSH Terms: conditions — Chikungunya Fever | interventions — Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Intervention Model Description: Prospective, comparator controled, randomized, double-blinded, interventional, safety study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects will receive two intramuscular injections on day 0 and 28 and one subcutaneous injection on day 0.
  Subjects randomized to verum will receive MV-CHIK intramuscularely on days 0 and 28 and placebo subcutaneously in the contralateral arm on day 0.
  Subjects randomized to the comparator will receive MMR-vaccine subcutaneously on day 0 and placebo (dummy injection) intramuscularely on days 0 and 28 in the contralateral arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MV-CHIK and Placebo (Experimental): Subjects will receive two injections on study day 0 and one injection on day 28.
  On both days they will receive a 5E+05 (+/- 0.5 log) TCID50 intramuscularly in the deltoid muscle of one arm.
  On day 0 they will receive a dummy injection of placebo (physiological saline) subcutaneously in the contralateral arm.
  Interventions: Biological: MV-CHIK
- MMR-vaccine and Placebo (Active Comparator): Subjects will receive two injections on study day 0 and one injection on day 28.
  On both days they will receive dummy injections of placebo (physiological saline) in the deltoid muscle of one arm.
  On day 0 they will receive MMR-vaccine subcutaneously in the contralateral arm.
  Interventions: Biological: MMR-vaccine

INTERVENTIONS:
Biological: MV-CHIK — Lyophilized, life attenuated, measles vectored Chikungunya vaccine; 5E+05 TCID50 (+/- 0.5 log) per dose
  Other Names: MV-CHIK vaccine; MV-CHIK/DP
  Arms: MV-CHIK and Placebo
Biological: MMR-vaccine — Lyophilized mixture of life attenuated Measles, Mumps, and Rubella viruses; 1000, 12500, and 1000, respectively, TCID50 per dose
  Other Names: MPR vaccine
  Arms: MMR-vaccine and Placebo

SUMMARY:
The clinical study primarily assesses the safety of MV-CHIK a new Chikungunya vaccine in a previously epidemic area in healthy volunteers. Secondarily, immune response and viremia will be assessed.

MV-CHIK will be compared to the commercially available MMR vaccine. 80% of the subjects will receive MV-CHIK; 20% will receive MMR vaccine.

DETAILED DESCRIPTION:
The clinical study to be conducted under this IND will assess the safety of MV-CHIK in a previously epidemic area (Puerto Rico).

A total of 100 healthy volunteers, 50 of whom are seropositive to Chikungunya at baseline and 50 of whom are seronegative, will be randomized in a 4:1 ratio to receive either MV-CHIK or the commercially available MMR vaccine in a double blinded fashion. Memory aids, to be completed by the volunteer at home, and the investigator at scheduled follow-up visits, will solicit symptoms of injection site reactions, fever, headache, malaise, joint and muscle pain. Acute phase reactants (C-reactive protein and ferritin) will be checked routinely throughout the study and at the discretion of the investigator in order to help determine if symptoms, particularly those referred to the joints, have an immunological basis.

This study will also evaluate the immune response in Chikungunya-exposed versus unexposed individuals by comparing neutralizing antibody titers at specific time points. Measles viremia will also be measured and compared between MV-CHIK and MMR recipients, and at three days after the second versus after the first dose. The relationship between measles viremia and the immune response to MV-CHIK will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥21 to ≤50 years on the day of enrollment.
2. Able to provide informed consent.
3. Available and accessible for the duration of the trial.
4. Able and willing to comply with all requirements of the study.
5. For female subjects, willing to practice a reliable form of contraception as specified in the protocol until five months after the second and final vaccination in accordance with recommendations following MMR vaccination.
6. Medical history and physical examination findings are considered normal or not clinically significant in the opinion of the Investigator.
7. Laboratory values are considered normal or not clinically significant in the opinion of the Investigator.
8. History of previous measles vaccination, either in childhood or as an adult if more than three months before participation in this study.

Exclusion Criteria:

1. Taking medication or other treatment for unresolved symptoms attributed to a previous chikungunya virus infection.
2. Prior receipt of any chikungunya or other alphavirus vaccine.
3. Recent infection, including suspected chikungunya (within 1 week prior to Screening Visit).
4. History of an allergic or anaphylactic reaction to any vaccine.
5. An allergic reaction other than allergic contact dermatitis to any component of either vaccine (i.e., neomycin, gelatin), or a current egg allergy. Volunteers with a childhood history of egg allergy who are able to tolerate egg in their diet now will not be excluded on this basis.
6. History of an immunosuppressive disorder (such as human immunodeficiency virus [HIV] infection, common variable immunodeficiency), chronic infection (such as chronic hepatitis B or C), autoimmune disease (such as rheumatoid arthritis, systemic lupus erythematosus [SLE], autoimmune thyroid disease) or any medical condition that, in the opinion of the Investigator, could lead to an atypical immune response to the vaccine.
7. History of moderate or severe non-traumatic arthritis or arthralgia within 3 months of the Screening Visit.
8. Recent (within 30 days), current or anticipated use of any immunosuppressive or immune modifying medication including corticosteroids (excluding nasal, ophthalmic, and other topical preparations).
9. Other vaccination or planned vaccination within 4 weeks of either study dose (seasonal influenza vaccine excepted).
10. Measles vaccination or booster within the last 3 months or planned during the clinical study.
11. Receipt or planned receipt of blood products including immunoglobulins within 120 days of the Screening Visit.
12. Pregnant or lactating or planning pregnancy during the trial.
13. Known alcohol or other substance abuse that in the opinion of the Investigator affects the ability or willingness of the participant to understand and comply with the study protocol.
14. Participation in another clinical study within the past 30 days in which the subject was exposed to an investigational product (pharmaceutical product or placebo or device) or planned concurrent participation in another clinical study during the study period.
15. Relevant history of any medical condition that, in the opinion of the Investigator, may interfere with the safety of the subject (volunteer) or aims of the study.
16. History of neoplastic disease (excluding successfully treated non-melanoma skin cancer or cervical intraepithelial neoplasia) within the past 5 years or a history of any hematological malignancy.
17. Behavioral or psychiatric disease or cognitive impairment that in the opinion of the Investigator affects the ability or willingness of the participant to understand and comply with the study protocol.
18. Non-consent to storage of blood specimens for future research.
19. Persons in direct relationship with the Sponsor or its contract service provider, the clinical research organization (CRO) or its subcontractors, the Investigator or study site staff. Direct relationship includes first degree relatives or dependents (children, spouse/partner, siblings or parents), as well as employees (site or Sponsor). Employees of the University of Puerto Rico not directly employed by the Clinical & Translational Research Center will not be excluded.
20. Any condition that would, in the opinion of the site Investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clemente Diaz, MD, Principal Investigator — University of Puerto Rico
Locations (1):
- University of Puerto Rico - Medical Sciences Campus, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MV-CHIK and Placebo: Subjects will receive two injections on study day 0 and one injection on day 28.
  On both days they will receive a 5E+05 (+/- 0.5 log) TCID50 intramuscularly in the deltoid muscle of one arm.
  On day 0 they will receive a dummy injection of placebo (physiological saline) subcutaneously in the contralateral arm.
  MV-CHIK: Lyophilized, life attenuated, measles vectored Chikungunya vaccine; 5E+05 TCID50 (+/- 0.5 log) per dose
- MMR-vaccine and Placebo: Subjects will receive two injections on study day 0 and one injection on day 28.
  On both days they will receive dummy injections of placebo (physiological saline) in the deltoid muscle of one arm.
  On day 0 they will receive MMR-vaccine subcutaneously in the contralateral arm.
  MMR-vaccine: Lyophilized mixture of life attenuated Measles, Mumps, and Rubella viruses; 1000, 12500, and 1000, respectively, TCID50 per dose
Period: Overall Study
Arm/Group | MV-CHIK and Placebo | MMR-vaccine and Placebo
Started | 26 (First subject signed ICF (MV-CHIK group)) | 8 (First subject signed ICF (MMR group))
Completed | 23 (End of Study Visit) | 7 (End of Study Visit)
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Population: MV-CHIK group: 12 seropositive, 14 seronegative subjects MMR-Placebo: 4 seropositive, 4 seronegative subjects
Groups:
- MV-CHIK-Placebo: 2 MV-CHIK injections (day 0+day 28); 1 Placebo injection (day 0)
- MMR-Placebo: 2 Placebo injections (day 0+day 28); 1 MMR injection (day 0)
- Total: Total of all reporting groups
Arm/Group | MV-CHIK-Placebo | MMR-Placebo | Total
Number analyzed (Participants) | 26 | 8 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 8 | 34
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (8.27) | 33.2 (8.27) | 33.2 (8.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 14
  Male | 15 | 5 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 8 | 34
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 26 | 8 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With AEs and Abnormal Lab Values, Vital Signs, and PE Findings
Description: Number of solicited and unsolicited adverse events and number of grade 2 and higher solicited and unsolicited adverse events including clinically significant abnormal safety laboratory results, vital signs, and physical examination findings in previously exposed versus unexposed individuals.
Time Frame: Throughout the whole study period (until day 392 after first dose)
Population: The intent-to-treat (ITT) population included all subjects who were randomized and received at least 1 dose of IVP. The ITT population was used for the safety analyses. Subjects were reported based on actual vaccine received.
Measure: Number; unit: subjects
Groups:
- MV-CHIK-Placebo/Seropositive: baseline seropositive cohort; received MV-CHIK-Placebo
- MV-CHIK-Placebo/Seronegative: baseline seronegative cohort; received MV-CHIK-Placebo
- MMR-Placebo/Seropositive: baseline seropositive cohort; received MMR-Placebo
- MMR-Placebo/Seronegative: baseline seronegative cohort; received MMR-Placebo
Arm/Group | MV-CHIK-Placebo/Seropositive | MV-CHIK-Placebo/Seronegative | MMR-Placebo/Seropositive | MMR-Placebo/Seronegative
Number analyzed (Participants) | 12 | 14 | 4 | 4
subjects
  All AEs | 11 | 13 | 4 | 4
  Severity: Severe | 0 | 2 | 0 | 1
  Severity: Moderate | 4 | 6 | 0 | 1
  Severity: Mild | 10 | 13 | 4 | 4
  IVP related AEs | 2 | 1 | 1 | 0
  (IVP Rel.AEs) Severity: Severe | 0 | 0 | 0 | 0
  (IVP Rel.AEs) Severity: Moderate | 1 | 0 | 0 | 0
  (IVP Rel.AEs) Severity: Mild | 1 | 1 | 1 | 0
  SAEs | 0 | 0 | 0 | 0

2. Secondary Outcome: Immunogenicity
Description: Immunogenicity on days 0, 28, 56, 168, 280, and at the end of the study measured as geometric mean titer (GMT) of neutralizing antibodies to chikungunya in previously exposed versus unexposed individuals.
Time Frame: Days 0, 28, 56, 168, 280, and 392
Population: The per protocol (PP) population was a subset of the ITT population that included subjects who received both doses of IVP, had at least 1 post-vaccination immunogenicity assessment, and did not experience a protocol deviation that could have affected their evaluation for immunogenicity. Protocol deviations that affected evaluation of immunogenicity were determined based on a blinded data review prior to database lock.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MV-CHIK-Placebo/Seropositive | MV-CHIK-Placebo/Seronegative | MMR-Placebo/Seropositive | MMR-Placebo/Seronegative
Number analyzed (Participants) | 11 | 14 | 4 | 3
Titer
  Day 0: number analyzed (Participants) | 11 | 12 | 4 | 3
  Day 0 | 1059.52 [762.0 to 1473.3] | 5.0 [3.6 to 6.9] | 1280.0 [740.9 to 2211.3] | 5.0 [2.7 to 9.4]
  Day 28: number analyzed (Participants) | 10 | 12 | 4 | 3
  Day 28 | 1290.19 [919.8 to 1809.8] | 17.82 [13.0 to 24.4] | 1280.0 [740.9 to 2211.3] | 5.0 [2.7 to 9.4]
  Day 56: number analyzed (Participants) | 11 | 12 | 4 | 3
  Day 56 | 1280.0 [920.5 to 1779.9] | 339.03 [247.3 to 464.9] | 1280.0 [740.9 to 2211.3] | 5.0 [2.7 to 9.4]
  Day 168: number analyzed (Participants) | 11 | 12 | 4 | 3
  Day 168 | 1280.0 [920.5 to 1779.9] | 63.5 [46.3 to 87.1] | 1280.0 [740.9 to 2211.3] | 5.0 [2.7 to 9.4]
  Day 280: number analyzed (Participants) | 10 | 12 | 4 | 2
  Day 280 | 1114.3 [792.2 to 1567.3] | 35.64 [26.0 to 48.9] | 1280.0 [740.9 to 2211.3] | 5.0 [2.5 to 10.2]
  End of Study: number analyzed (Participants) | 10 | 12 | 4 | 3
  End of Study | 1280.00 [907.0 to 1806] | 29.97 [21.9 to 41.1] | 1280.00 [740.9 to 2211.3] | 5.00 [2.7 to 9.4]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were monitored throughout the study. Under protocol versions 1.0 and 2.0, nonserious AEs were recorded from the time a subject signed the ICF, Under protocol version 3.0, nonserious AEs were recorded from the time a subject received their first vaccination on Day 0 through the last follow-up visit on Day 392 (±10 days).
Description: Adverse event of special interest:The AESI for this study, persistent joint pain, was defined as nontraumatic joint pain or stiffness that persisted for more than 24 hours or was associated with objective findings of effusion or soft tissue swelling.
Arm/Group | MV-CHIK-Placebo/Seronegative | MV-CHIK-Placebo/Seropositive | MMR-Placebo/Seropositive | MMR-Placebo/Seronegative
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 11/12 | 13/14 | 4/4 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MV-CHIK-Placebo/Seronegative (N=12) | MV-CHIK-Placebo/Seropositive (N=14) | MMR-Placebo/Seropositive (N=4) | MMR-Placebo/Seronegative (N=4)
Infections and infestations (Infections and infestations) | 3 | 7 | 4 | 3
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 6 | 4 | 1 | 2
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 4 | 2 | 0 | 1
Nervous system disorders (Nervous system disorders) | 3 | 1 | 1 | 1
Respiratory, thoracic, mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 0
Gastrointestinal disorders (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 1
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 | 4 | 0 | 0
Renal and urinary disorders (Renal and urinary disorders) | 0 | 4 | 0 | 0
Cardiac disorders (Cardiac disorders) | 0 | 0 | 2 | 0
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Vascular disorders (Vascular disorders) | 2 | 0 | 0 | 0
Investigations (Investigations) | 1 | 0 | 0 | 0
Psychiatric disorders (Psychiatric disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT03101111/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT03101111/SAP_001.pdf